CLINICAL TRIAL: NCT05794516
Title: A Single Ascending Dose (SAD) Study to Evaluate the Safety and Pharmacokinetics (PK) of ZB004 in Healthy Volunteers
Brief Title: A Safety and Pharmacokinetics Study of ZB004 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zenas BioPharma (USA), LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZB004-01-001
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZB004 (Experimental)
  Interventions: Drug: ZB004
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZB004 — ZB004 single doses administered subcutaneously as solution
  Arms: ZB004
Drug: Placebo — Placebo single doses administered subcutaneously as solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of single-ascending doses of ZB004.

DETAILED DESCRIPTION:
Up to approximately 40 healthy volunteers across 5 cohorts randomized to receive ZB004 or placebo as single doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female participants 18 to 55 years of age.
* Body weight ≥ 50 kg for male participants and ≥ 45 kg for female participants; body mass index of 18 to 35 kg/m^2 for both male and female participants.
* Considered in good health as determined by the Investigator.
* Female participants of child-bearing potential must agree to abstinence or use an highly effective form of contraception. Female participants must also refrain from donation of eggs from the signing of the informed consent to 6 months after receiving their dose of study drug.
* Male participants must be surgically sterile or agree to use effective contraception. Male participants must also agree not to donate sperm from the signing of the informed consent to 6 months after the last scheduled dose of the study drug.
* Willing and able to understand the characteristics and purposes of the study, including possible risks involved, and willing to comply with all the study requirements and provide written informed consent for the study.

Exclusion Criteria:

* Surgery within 4 weeks before Screening or planned surgery during the clinical study.
* Use of prescription medications, biological products, or other medicines within 2 weeks before Study Day 1 or 5 half-lives of the product, whichever is greater. Use of over-the-counter medications or vitamins/dietary supplements within 7 days of dosing unless considered by the Investigator to not pose a risk or impact the study results.
* Clinically significant ECG abnormality.
* Positive for HIV, active hepatitis C or B, Covid-19 virus, tuberculosis.
* Bacteria, viruses, systemic fungi, parasites, or other opportunistic infections within 30 days before Study Day 1.
* History of drug abuse in the previous 12 months before Screening, or positive for urine drug Screening (Day -28 to Day -1).
* Donated blood (including component blood) or lost > 400 mL within 3 months before Screening or received a transfusion within 3 months of Screening.
* History of relevant allergies (including allergy to any murine or human-derived protein or immunoglobulin products, rubber or latex, or other allergies that in the opinion of the Investigator make inclusion in the study inappropriate).
* Average daily smoking > 10 cigarettes/day (or equivalent) within 6 months of Screening.
* Consume > 14 standard units of alcohol per week (1 standard unit is equivalent to approximately 360 mL of beer, 45 mL of spirits with 40% alcohol, or 150 mL of wine) or a positive alcohol breath test on Day -1.
* Any disease that might interfere with the safety evaluation of the investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) to evaluate Safety and Tolerability of ZB004 | Day 1 through Day 99

SECONDARY OUTCOMES:
Number of participants with treatment-emergent serious adverse events (SAEs) | Day 1 through Day 99
Number of participants with laboratory abnormalities | Day 1 through Day 99
Number of participants with Electrocardiogram (ECG) abnormalities | Day 1 through Day 99
Maximum observed serum concentration (Cmax) | Day 1 through Day 99
Time for Cmax (Tmax) | Day 1 through Day 99
Area under the concentration-time curve from Time 0 extrapolated to infinity (AUCinf) | Day 1 through Day 99
AUC from time 0 to the last quantifiable concentration (AUClast) | Day 1 through Day 99
Terminal half-life (t½) | Day 1 through Day 99
Apparent clearance following extravascular dosing (CL/F) | Day 1 through Day 99
Apparent volume of distribution following extravascular administration (Vz/F) | Day 1 through Day 99

CONTACTS AND LOCATIONS:
Locations (1):
- NZCR New Zealand Clinical Research, Christchurch, New Zealand